CLINICAL TRIAL: NCT01520428
Title: Interventions to Prevent Adolescents With Type 1 Diabetes From Long-term Complications. A Multicenter Randomized Controlled Trial
Brief Title: Interventions to Prevent Adolescents With Type 1 Diabetes From Long-term Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: National Bank of Austria (Other Government)
Responsible Party: Principal Investigator, Rami-Merhar, Birgit, Univ. Prof. Dr. Med. MBA, Univ.Prof.Dr.Med.MBA, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ÖNB13686
Record Dates: First submitted 2012-01-19; First posted 2012-01-30 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing, CBT and E-mail support (Active Comparator)
  Interventions: Behavioral: Motivational Interviewing, CBT and E-mail support
- E-Mail-support (Active Comparator)
  Interventions: Behavioral: Motivational Interviewing, CBT and E-mail support

INTERVENTIONS:
Behavioral: Motivational Interviewing, CBT and E-mail support — Motivational Interviewing, elements of Cognitive Behaviour Therapy and E-mail support
  Other Names: Motivational Interviewing, Cognitive Behaviour Therapy, Diabetes mellitus type 1, children, adolescents

SUMMARY:
The purpose of this study is to evaluate the effectiveness of diabetes management training combined with the method of Motivational Interviewing with elements of Cognitive Behaviour Therapy and E-mail support in the treatment of type 1 diabetes in adolescents (age range 13-20 years) compared to a control group. The investigators assess motivational changes and effects on metabolic control.

DETAILED DESCRIPTION:
Diabetes mellitus type1 requires lifelong insulin substitution, aiming at near normal glycaemia. Insufficient metabolic control (HbA1c > 8 %) leads to micro and macro- vascular complications. Especially in adolescence a lack of compliance leads to deteriorated metabolic control. Motivational factors play a pivotal role in this age-group, however they have neither been studied so far nor considered in interventions with diabetes patients.

Therefore, the aim of this study is to evaluate in a multi-centred randomized controlled trial the effectiveness of diabetes management training with the method of Motivational Interviewing with elements of Cognitive Behaviour Therapy and E-mail support.

Sixty adolescents within the age group of 13-20 years and HbA1c levels > 8 % will - after a refresher course in diabetes education - be involved to 2-weekly individual interventions sessions including motivational interviewing and CBT-modules with a psychologist and weekly e-mail support for a period of six month in order to improve HbA1c levels, self- efficacy in diabetes management and general quality of life.

As control group sixty adolescents within the age group of 13-20 years and HbA1c levels > 8 will - after a refresher course in diabetes education - get treatment as usual, including routine medical support visits, unspecific psychological consultations and unspecific e-mail support to match with the intervention group for time bonus.

We assess motivational changes and effects on metabolic control (HbA1c) and define the predictors of positive effects on glycaemic control.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, type1
* HbA1c>8
* 1 year of diagnosis
* Access to Internet available

Exclusion Criteria:

* N/A

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
HbA1C | after 8 months
  Metabolic control

SECONDARY OUTCOMES:
Predictors of positive effects on glycaemic control | after 6 months and after 12 months
Motivational changes | after 6 months and 12 months
HbA1c | after 12 months
  Metabolic control

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Rami-Merhar, MD, Uni Prof, Principal Investigator — Medical University of Vienna, Dep. of Pediatrics and Adolescent Medicine
Locations (1):
- Medical University of Vienna, Vienna, Austria